CLINICAL TRIAL: NCT03696095
Title: Continuous Infusion vs. Programmed Intermittent Bolus of Ropivacaine Through Peri-neural Femoral Nerve Catheter After Total Knee Arthroplasty: Impact on Analgesia Quality and Motor Block Frequency.
Brief Title: Local Anesthetic Automated Intermittent Administration vs. Continuous Infusion Via Femoral Nerve Block.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: J P Lecoq (Other)
Responsible Party: Sponsor-Investigator, J P Lecoq, MD, University of Liege
Organization: University of Liege (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-000822-70
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Pain; Postoperative Complications
Keywords: total knee arthroplasty; postoperative pain; programmed intermittent bolus; Continuous femoral nerve block
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continous infusion ropivacaine (Active Comparator): Continuous infusion via peri-neural femoral nerve catheter of Ropivacaine Hcl 0.2% Inj Bag 200Ml (CI mode) at rate of 6ml/h + patient controlled bolus of 3ml ...
  Interventions: Drug: Ropivacaine Hcl 0.2% Inj Bag 200Ml (CI mode)
- PIB ropivacaine (Experimental): Programmed intermittent bolus of Ropivacaine Hcl 0.2% Inj Bag 200Ml (PIB mode) : 6ml each 60min + patient controlled bolus 3ml ...
  Interventions: Drug: Ropivacaine Hcl 0.2% Inj Bag 200Ml (PIB mode)

INTERVENTIONS:
Drug: Ropivacaine Hcl 0.2% Inj Bag 200Ml (PIB mode) — programmed intermittent bolus 5ml each one hour.
  Other Names: PIB
  Arms: PIB ropivacaine
Drug: Ropivacaine Hcl 0.2% Inj Bag 200Ml (CI mode) — continuous infusion 6ml/h
  Other Names: Continuous infusion
  Arms: Continous infusion ropivacaine

SUMMARY:
This study evaluates the impact of local anesthetic administration regiment through peri-neural femoral nerve catheter on pain and motor block frequency, after total knee arthroplasty.

DETAILED DESCRIPTION:
This study evaluates the impact of local anesthetic administration regiment through peri-neural femoral nerve catheter on pain and motor block frequency, after total knee arthroplasty. One group of patients will receive automated intermittent bolus, while the others will get a continuous infusion. In both cases, patients will be able to administer supplementary auto-bolus if required.

ELIGIBILITY:
Inclusion Criteria:

* admitted for unilateral primary total knee arthroplasty.

Exclusion Criteria:

* ASA score > 3
* BMI > 40
* refusal of loco-regional technique.
* psychiatric disease.
* inability to understand/ use the Local anesthetic delivery pump.
* local anesthetic allergy,
* porphyry,
* uncontrolled epilepsy,
* severe cardiac arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Frequency of unplanned analgesia interventions. | up to 72 hours after surgery
  Composite criteria including the frequency of unplanned analgesia interventions administered by the patient, or paramedical and medical staff, and by extenstion the total amount of opioids (in milligrams equivalent morphine) and local anesthetics (in milligrams) received in post-operative period.

SECONDARY OUTCOMES:
Pain difference | up to 72 hours after surgery
  Pain difference accessed by Numeric Pain Rating Scale (0-10), twice a day, at rest and on movement.
Motor block frequency | up to 72 hours after surgery
  Accessed by physiotherapist twice a day, by testing the Quadriceps muscle.
Mobilization quality during physiotherapy sessions. | up to 72 hours after surgery
  accessed by physiotherapist, ability to walk with or without help, take stairs, and flex and extend knee (comparatively to the opposite knee).
local anesthesia technique related complications | until catheter removal 48 hours after surgery
  rate of complications including: hematoma, infection, catheter dislodgement or breakage, allergic events.

CONTACTS AND LOCATIONS:
Overall Officials: Annis Orfi, Principal Investigator — University of Liege
Locations (1):
- CHU Liege, Liège, Belgium